CLINICAL TRIAL: NCT03282838
Title: Open-Label, Three Way, Randomized, Single Dose Crossover Study Comparing Bioavailability of DFN-15 Oral Solution Under Fasting Conditions vs Comparator Under Fed Conditions and to Determine Food Effect of DFN-15 in Healthy Adult Subjects
Brief Title: Study on the Pharmacokinetics (PK) of DFN-15 vs Comparator and Food-effect on DFN-15 PK in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DFN-15-CD-008
Record Dates: First submitted 2017-08-17; First posted 2017-09-14 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DFN-15 (fasted) (Experimental)
  Interventions: Drug: DFN-15 (fasted)
- DFN-15 (fed) (Experimental)
  Interventions: Drug: DFN-15 (fed)
- Comparator (fed) (Experimental)
  Interventions: Drug: Comparator Celebrex® (fed)

INTERVENTIONS:
Drug: DFN-15 (fasted) — DFN-15 administered to fasted subjects
  Arms: DFN-15 (fasted)
Drug: DFN-15 (fed) — DFN-15 administered to fed subjects
  Arms: DFN-15 (fed)
Drug: Comparator Celebrex® (fed) — Comparator (Celebrex®) administered to fed subjects
  Arms: Comparator (fed)

SUMMARY:
An Open-Label, Three-Way Randomized, Single Dose Crossover Study Comparing Bioavailability of DFN-15 under fasting conditions versus Comparator under fed conditions and to determine food-effect of DFN-15 in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female 19-55 years of age, inclusive, at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
* Females of childbearing potential: must either be sexually inactive (abstinent) for 30 days prior to the first dose and throughout the study or be using birth control method; Female subjects of non-childbearing potential and must have undergone sterilization procedures or be postmenopausal for at least 1 year prior
* Male subject must agree to use contraception or abstain during the study until 90 days beyond the last dose of study drug.
* Understands the study procedures in the informed consent form (ICF), and willing and able to comply with the protocol.

Exclusion Criteria:

* History or presence of hypersensitivity or idiosyncratic reaction to celecoxib, sulfonamides, aspirin or other NSAIDs or related compounds
* History or presence of clinically significant medical or psychiatric condition or disease
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* liver enzyme tests greater than the upper limit of normal at screening
* Estimated creatinine clearance <90 mL/minute at screening
* History or presence of alcoholism
* History or presence of bilateral pedal edema or generalized edema or fluid retention
* Female subjects who are pregnant or lactating or actively trying to conceive
* Positive urine drug or alcohol results at screening or check-in
* Positive cotinine at screening
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)
* Seated blood pressure is less than 90/60 mmHg or greater than 140/90 mmHg at screening
* Seated heart rate is lower than 45 bpm or higher than 100 bpm at screening
* Has been on a diet incompatible with the on-study diet
* Unable to refrain from or anticipates the use of prohibited medications
* Donation of blood or significant blood loss within 56 days prior to the first dose of study drug; plasma donation within 7 days prior to the first dose of study drug
* Participation in another clinical trial within 28 days prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
DFN-15 maximum plasma concentration (Cmax) | Up to 72 hours
DFN-15 area under the curve (AUC) 0-t | Up to 72 hours
DFN-15 area under the curve (AUC) 0-inf | Up to 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided